CLINICAL TRIAL: NCT04147975
Title: Assessment of Assay for Rapid Identification of Bloodstream Infections From Whole Blood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HelixBind, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20031
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Bacteremia; Candidemia
MeSH Terms: conditions — Bacteremia; Candidemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients Suspected of Bloodstream Infection: No intervention(s) to be administered.
  Interventions: Diagnostic Test: RaPID/BSI Test

INTERVENTIONS:
Diagnostic Test: RaPID/BSI Test — RaPID/BSI Test

SUMMARY:
The purpose of this study is to assess the effectiveness of RaPID/BSI by testing its performance compared to blood cultures collected prospectively from consented subjects.

ELIGIBILITY:
Inclusion Criteria:

* Determined to have a positive blood culture.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who are culture positive for bacterial or fungal bloodstream infection.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity compared to Blood Culture (comparator method) | Up to 24 hours following blood collection
  The primary endpoint of sensitivity (detection of on panel pathogen) and specificity will be determined by comparing blood culture results with the RaPID/BSI results from the prospective clinical specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- HelixBind Inc., Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No